CLINICAL TRIAL: NCT06123364
Title: The Effects of Extracorporeal Magnetic Innervation in Combination With Mirabegron in the Treatment of Urinary Frequency, Urgency and Urge Incontinence
Brief Title: Extracorporeal Magnetic Innervation in Combination With Mirabegron in the Treatment of Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serdinsek Tamara (Other)
Responsible Party: Sponsor-Investigator, Serdinsek Tamara, Assistant professor, MD, PhD, University Medical Centre Maribor
Organization: University Medical Centre Maribor (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRP-2018/01-06
Record Dates: First submitted 2023-10-29; First posted 2023-11-08 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome
Keywords: overactive bladder; urinary urge incontinence; mirabegron; magnetic stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 study groups, namely one group will receive actual electromagnetic stimulation, and the other group will receive placebo stimulation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment arm (Active Comparator): Patients in this study arm will receive 50 mg of mirabegron daily in the form of tablets, which is used to treat OAB according to current treatment guidelines. Additionally they will twice a week receive an actual extracorporeal electromagnetic stimulation in the duration of 20 minutes, for 8 weeks.
  Interventions: Drug: mirabegron 50 mg daily; Device: Extracorporeal magnetic innervation (active treatment)
- Sham treatment arm (Sham Comparator): Patients in this study arm will receive 50 mg of mirabegron daily in the form of tablets, which is used to treat OAB according to current treatment guidelines. Additionally they will twice a week receive a sham extracorporeal electromagnetic stimulation in the duration of 20 minutes, for 8 weeks.
  Interventions: Drug: mirabegron 50 mg daily; Device: Extracorporeal magnetic innervation (sham treatment)

INTERVENTIONS:
Drug: mirabegron 50 mg daily — Patients in both study groups will receive 50 mg of mirabegron daily in the form of tablets, which is used to treat OAB according to current treatment guidelines.
Device: Extracorporeal magnetic innervation (active treatment) — Patients will twice a week receive extracorporeal electromagnetic stimulation in the duration of 20 minutes. Patients will be randomized into 2 study groups, namely one group will receive actual electromagnetic stimulation, and the other group will receive sham stimulation.
  Arms: Active treatment arm
Device: Extracorporeal magnetic innervation (sham treatment) — Patients will twice a week receive extracorporeal electromagnetic stimulation in the duration of 20 minutes. Patients will be randomized into 2 study groups, namely one group will receive actual electromagnetic stimulation, and the other group will receive placebo stimulation.
  Arms: Sham treatment arm

SUMMARY:
The goal of this clinical trial is to learn about impact of extracorporeal electromagnetic stimulation in addition to medical treatment with mirabegron on the treatment of overactive bladder (OAB). The study will include female patients, aged between 30 and 80, with signs of OAB, including urinary frequency, urgency and urinary urgency incontinence.

The main questions it aims to answer are:

* Does the addition of extracorporeal electromagnetic stimulation to medical treatment with mirabegron influence the urinary urgency incontinent or frequency?
* Does the addition of extracorporeal electromagnetic stimulation to medical treatment with mirabegron influence the urine flow or post-void residual volume?
* Does the addition of extracorporeal electromagnetic stimulation to medical treatment with mirabegron influence the patients' quality of life.

Participants will:

* receive 50 mg of mirabegron daily in the form of tablets, which is used to treat OAB according to current treatment guidelines.
* Twice a week receive extracorporeal electromagnetic stimulation in the duration of 20 minutes. The patients will be divided into 2 groups, namely one group will receive actual electromagnetic stimulation, and the other group will receive placebo stimulation.
* Have a urogynecological examination, with ultrasound measurements of the remaining urine in the bladder and determination of the thickness of the bladder wall, as well as a uroflow examination, after 4 and 8 weeks of treatment.
* Have to to submit urine for laboratory tests and to fill out questionnaires regarding participants' symptoms, after 4 and 8 weeks of treatment.

Researchers will compare both study groups to see if the addition of extracorporeal electromagnetic stimulation has influence on the research questions stated above.

DETAILED DESCRIPTION:
In this study the investigators are studying the impact of extracorporeal electromagnetic stimulation on the treatment of overactive bladder (OAB).

For the research, the investigators will gather participants' basic demographic information (age, co-morbidities, etc.), results of uro-gynecological examinations (gynecological and transabdominal ultrasound, uroflow, urinalysis) and the results of different questionnaires, which will be filled out by the participants, describing the burden of the investigated disease and the impact on quality of life.

The research will last 8 weeks. Before the start of the research, participants will submit a urine sample to rule out a urinary tract infection and determine baseline laboratory parameters in the urine. Participants will then receive 50 mg of mirabegron daily in the form of tablets, which is used to treat OAB according to current treatment guidelines. Twice a week participants will come to the Department of General Gynecology and Gynecological Urology, Clinic of Gynecology and Perinatology, UMC Maribor, where the investigators will additionally perform extracorporeal electromagnetic stimulation for the treatment of OAB. These treatments will last 20 minutes each time. The patients will be divided into 2 groups, namely one group will receive actual electromagnetic stimulation, and the other group will receive placebo stimulation.

At the beginning of the research and after 4 and 8 weeks, the investigators will perform a uro-gynecological examination, with ultrasound measurements of the remaining urine in the bladder and determination of the thickness of the bladder wall, as well as a uroflow examination. It will be necessary for the participants to submit urine for laboratory tests and to fill out questionnaires regarding OAB symptoms.

Based on the safety profile of mirabegron and extracorporeal electromagnetic stimulation, the investigators do not expect any serious side effects. The investigators anticipate that there will be a reduction in the symptoms caused by the overactive bladder. In the event of a serious adverse event, participants can contact the on-call gynecologist or on-call urologist at UMC Maribor, who are available 24 hours a day.

In the research, the participants' personal data will remain undisclosed, as the investigators will lead each participant under a random number during data processing, and will also display the results in the form of an average for the entire group of participants, so that it will not be possible to draw conclusions about participants' identity based on the results. Participation in the research is voluntary, and participants can stop participating at any stage of the research.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Age between 30 and 80 years
* Signs of OAB (including urinary frequency, urgency and urinary urgency incontinence)

Exclusion Criteria:

* Positive urine culture
* Treatment with anticholinergics or mirabegron in the last 3 months
* Physiotherapy treatment of the pelvic floor muscles (e.g. pelvic floor exercises, electrical stimulation, etc.) in the last 3 months
* Stress incontinence
* Pelvic malignancies
* Pregnancy
* Cardiac pacemaker, implantable cardiac defibrillator
* Electronic device or metallic implant applied to areas between the lumbar region and lower extremities

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in the rate of urgency incontinence episodes | From enrollment to the end of treatment at 8 weeks
  The investigators will monitor the rate of urgency incontinence episodes at the enrollment and throughout the study to detect a possible urgency incontinence rate change.

SECONDARY OUTCOMES:
Change in Incontinence Quality of Life Questionnaire (I-QOL) Score | From enrollment to the end of treatment at 8 weeks
  The investigators will monitor the change in Incontinence Quality of Life Questionnaire (I-QOL) Score at the enrollment and throughout the study to detect a possible improvement in quality of life. The score rage is from values 0 to 100, where higher scores mean a better outcome.
Change in Incontinence Impact Questionnaire - short form (IIQ-7) Score | From enrollment to the end of treatment at 8 weeks
  The investigators will monitor the change in Incontinence Impact Questionnaire - short form (IIQ-7) Score at the enrollment and throughout the study to detect a possible improvement in quality of life. The score rage is from values 0 to 100, where lower scores mean a better outcome.
Change in Urogenital Distress Inventory - short form (UDI-6) Score | From enrollment to the end of treatment at 8 weeks
  The investigators will monitor the change in Urogenital Distress Inventory - short form (UDI-6) Score at the enrollment and throughout the study to detect a possible improvement in quality of life. The score rage is from values 0 to 100, where lower scores mean a better outcome.
Change in Patient Perception of Intensity of Urgency Scale (PPIUS) | From enrollment to the end of treatment at 8 weeks
  The investigators will monitor the change in Patient Perception of Intensity of Urgency Scale (PPIUS) at the enrollment and throughout the study to detect a possible improvement in quality of life. The score rage is from values 0 to 4, where lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Igor But, MD, PhD, Study Director — University Medical Centre Maribor
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia